CLINICAL TRIAL: NCT04323254
Title: The Language of Sleepiness
Brief Title: Language of Sleepiness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, San Diego (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Bernie.Sunwoo, Associate Professor of Medicine, University of California, San Diego
Other Study IDs: 190489
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Sleep; Sleep Disorder; Sleepiness
MeSH Terms: conditions — Sleep Wake Disorders; Sleepiness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Subjects will complete an electronic consent form and then fill out questionnaires on a tablet computer. The answers to the questions will be recorded to a secure electronic database, along with the results of a clinical overnight sleep study performed separately from this research study (this research study will not perform any overnight visits). After the overnight study diagnosis researchers will see which answers are most commonly given in association with each diagnosis. In addition, we will assess to what extent the sleep disorder impacts the patient's perception of his/her quality of life.

DETAILED DESCRIPTION:
Research questionnaires will be given along with the clinical intake form to all patients who are interested in participating in our study. Subjects will complete an electronic consent form and then proceed to questionnaires on a tablet computer (outlined below). The answers to the questions will be recorded to a secure electronic database, REDCap, along with the results of the overnight sleep study (when available). For the initial analysis, we will determine the sleep diagnosis and see which descriptors are most commonly used in association with each diagnosis. In addition, we will assess to what extent the sleep disorder impacts the patient's perception of his/her quality of life. These analyses will be simple correlations for the linear scales and unpaired t-tests to compare different diagnoses.

REDCap REDCap, is a password-protected secure web application that we will use to build and manage our study database. REDCap is a HIPAA-compliant environment. Subjects will have a coded study identifier associated with their research documents and questionnaires. Only key personnel on this study will have access to the study database.

Questionnaires:

* Work Productivity Impairement Questionnaire-The questionnaire assesses how much sleepiness has impacted the subject's ability to work.
* Language of Sleepiness Questionniare-The questionnaire will capture what descriptors those with sleep issues use prior to their sleep consulation.
* San Diego Wisdom Scale (SD-WISE) - The questionnaire assesses subject's wisdom scores.
* Functional Outcomes of Sleep Questionnaire - The questionnaire is a subjective measure of sleepiness and quality of life.
* Beck Depression Index II - The questionnaire assesses mental health (i.e. depression).

Study Visit Patients that elect to participate in the study will be consented in either the sleep clinic conference room or sleep clinic exam room. Subjects will then complete the questionnaires on a tablet. The research documents and questionnaires will be hosted on REDCap, a secure electronic database. For participants who are not comfortable with the electronic format, we will provide paper copies of the questionnaires and enter their data manually into REDCap.

The total study time is estimated to be <20 minutes, which includes the consent process. Administration of the questionnaires should take 5-7 minutes. These activities will be completed before the subject's sleep consultation.

After Study Visit:

We will access subjects' medical records to document their vitals, age, race/ethnicity, height, weight, date of birth, phone number, medications, medical and surgical history, alcohol history, illicit drug including cannabidiol, allergies, and Epworth Sleepiness Scale (ESS) value from the day of their study visit (i.e. first sleep consultation appointment). We will also collect data from their sleep study. If the subject completes a Home Sleep Test the following will be obtained: time to bed, wake time, apnea hypopnea index (AHI), apnea index (AI), hypopnea index (HI), obstructive apnea index (OAI), central apnea index (CAI), mixed apnea index (MAI), Cheyne - Stokes respiration, oxygen desaturation index (ODI), oxygen saturation, # of breaths, and pulse.

ELIGIBILITY:
Inclusion Criteria:

1. Total participants: 200 (UCSD only)
2. Ages: 18 - 89
3. Gender: Men and Women
4. Ethnic background: All

We will not recruit vulnerable patient groups.

Exclusion Criteria:

1. Prior Sleep consultation
2. Prisoners
3. Cognitive impairment, unable to provide consent, or unable to carry out research procedures

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients new to the UCSD Pulmonary and Sleep Clinic with no prior sleep consultations.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-03-23 (Actual); Primary Completion 2021-03-23 (Estimated); Study Completion 2021-03-23 (Estimated)

PRIMARY OUTCOMES:
Language of Sleepiness Questionniare | 5 minutes
  The questionnaire will capture what descriptors those with sleep issues use prior to their sleep consulation. Subjects will choose the best descriptors of their sleeping problem and rank the top five of them in order (under the word Rank in the Table). For the top three descriptors that they chose, they will rank them on a scale of 1-10 in severity (1= minor problem, 10=major problem).

SECONDARY OUTCOMES:
Work Productivity Impairement Questionnaire | 5 minutes
  The questionnaire assesses how much sleepiness has impacted the subject's ability to work. Subject will report how many hours they work and how many of those hours are affected by sleepiness. Subjects will then be asked about how much sleepiness or tiredness affected their productivity while working by ranking at which percentage of their usual productivity were they working in the last 30 days despite sleepiness/tiredness (0% = completely unable to perform work, 100% = Productivity not at all affected).
San Diego Wisdom Scale (SD-WISE) | 5 minutes
  The questionnaire assesses subject's wisdom scores on a scale of 1-5 within 6 categories: Decisiveness, Emotional Regulation, Self-Reflection, Pro-Social Behaviors, and Social Advising. Higher scores indicate higher levels of wisdom in each respective category.
Functional Outcomes of Sleep Questionnaire | 5 minutes
  The questionnaire is a subjective measure of sleepiness and quality of life. The score range is 0-28 points, with higher scores indicating greater insomnia severity. The suggested guidelines for score interpretation is 0 -7 for no clinically significant insomnia, 8-14 for subthreshold insomnia, 15-21 for clinical insomnia (moderate severity), and 22-28 for clinical insomnia (severe).
Beck Depression Index II | 5 minutes
  The questionnaire assesses mental health (i.e. depression). Each of the 21 items are given weighted values corresponding to a symptom of depression and summed to give a single score. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.

CONTACTS AND LOCATIONS:
Overall Officials: Bernie Sunwoo, MBBS, Principal Investigator — Faculty
Locations (2):
- United States (2):
  - UCSD Health - Pulmonary and Sleep Clinic, La Jolla, California
  - Altman Clinical and Translational Research Institute, San Diego, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jordan AS, McSharry DG, Malhotra A. Adult obstructive sleep apnoea. Lancet. 2014 Feb 22;383(9918):736-47. doi: 10.1016/S0140-6736(13)60734-5. Epub 2013 Aug 2. PMID 23910433
- [Background] Peppard PE, Young T, Barnet JH, Palta M, Hagen EW, Hla KM. Increased prevalence of sleep-disordered breathing in adults. Am J Epidemiol. 2013 May 1;177(9):1006-14. doi: 10.1093/aje/kws342. Epub 2013 Apr 14. PMID 23589584
- [Background] Heinzer R, Vat S, Marques-Vidal P, Marti-Soler H, Andries D, Tobback N, Mooser V, Preisig M, Malhotra A, Waeber G, Vollenweider P, Tafti M, Haba-Rubio J. Prevalence of sleep-disordered breathing in the general population: the HypnoLaus study. Lancet Respir Med. 2015 Apr;3(4):310-8. doi: 10.1016/S2213-2600(15)00043-0. Epub 2015 Feb 12. PMID 25682233
- [Background] Hirsch Allen AJM, Bansback N, Ayas NT. The effect of OSA on work disability and work-related injuries. Chest. 2015 May;147(5):1422-1428. doi: 10.1378/chest.14-1949. PMID 25940253
- [Background] Weaver TE, Maislin G, Dinges DF, Bloxham T, George CF, Greenberg H, Kader G, Mahowald M, Younger J, Pack AI. Relationship between hours of CPAP use and achieving normal levels of sleepiness and daily functioning. Sleep. 2007 Jun;30(6):711-9. doi: 10.1093/sleep/30.6.711. PMID 17580592
- [Background] Daurat A, Ricarrere M, Tiberge M. Decision making is affected in obstructive sleep apnoea syndrome. J Neuropsychol. 2013 Mar;7(1):139-44. doi: 10.1111/j.1748-6653.2012.02039.x. Epub 2012 Oct 23. PMID 23088593